CLINICAL TRIAL: NCT02177396
Title: A Prospective Randomized Open-Label Blinded End Point (PROBE) Trial Comparing MICARDIS® (Telmisartan) (80 mg QD) and Valsartan (80 mg QD) in Patients With Mild-to-Moderate Hypertension Using Ambulatory Blood Pressure Monitoring.
Brief Title: MICARDIS® and Valsartan in Patients With Mild-to-Moderate Hypertension Using Ambulatory Blood Pressure Monitoring
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 502.256
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Valsartan

ARMS (2):
- Telmisartan (Experimental)
  Interventions: Drug: Telmisartan; Drug: Placebo
- Valsartan (Active Comparator)
  Interventions: Drug: Valsartan; Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan
  Arms: Telmisartan
Drug: Valsartan
  Arms: Valsartan
Drug: Placebo

SUMMARY:
The primary aim of the trial was to compare the effect of telmisartan and valsartan in lowering ambulatory diastolic and/or systolic blood pressure in the last six hours of the dosing interval. Secondary variables included changes from baseline in diastolic and systolic blood pressures during other times during the 24-hour ABPM profile, changes from baseline in seated trough diastolic and systolic blood pressures as measured by manual cuff, and responder rates. Assessment of safety was also considered. Adverse events and use of concomitant therapies were monitored at each study visit. Blood pressure and heart rate were collected at each visit. Physical examination, electrocardiograms (ECG) and laboratory tests were completed during the trial as well.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate hypertension defined as mean seated diastolic blood pressure measurement of ≥ 95 mm Hg and ≤ 114 mm Hg, measured by manual cuff sphygmomanometer, on the last visit (Visit 6) of the four-week placebo run-in period (baseline BP)
* Mean seated systolic blood pressure ≥ 140 mm Hg and ≤ 200 mm Hg, measured by manual cuff at Visit 6 (baseline BP)
* A 24-hour mean ABPM measurement of ≥ 130/85 mm Hg evaluated at Visit 7 (baseline ABPM)
* Age 18 or older
* Ability to provide written informed consent

Exclusion Criteria:

* Pre-menopausal women (last menstruation ≤ 1 year prior to start of screening):

  * Who are not surgically sterile (hysterectomy, tubal ligation)
  * Who are NOT practicing acceptable means of birth control or who do NOT plan to continue using an acceptable method throughout the study. Acceptable methods of birth control include IUD (intrauterine device), oral, implantable or injectable contraceptives
* Any woman:

  * Who has a positive serum pregnancy test at screening (Visit 1) or baseline (Visit 7)
  * Who is nursing
* Hepatic and/or renal dysfunction as defined by the following laboratory parameters

  * SGPT (ALT) (serum glutamate pyruvate transaminase) or SGOT (AST) (serum glutamate oxaloacetate transaminase) greater than two times the upper limit of normal
  * Serum creatinine > 2.3 mg/dL
* At screening (Visit 1): clinically relevant sodium depletion, hyperkalemia, or hypokalemia
* Known or suspected secondary hypertension
* Bilateral renal artery stenosis; renal artery stenosis in a solitary kidney; post-renal transplant patients, presence of only one functioning kidney
* Congestive heart failure (NYHA (New York Heart Association) functional class CHF (congestive heart failure) III-IV
* Unstable angina within the past three months
* Stroke within the past six months
* Myocardial infarction or cardiac surgery within the past three months
* PTCA (percutaneous transluminal coronary angioplasty) within the past three months
* History of angioedema
* Sustained ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the investigator
* Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of the aortic or mitral valve
* Administration of digoxin or other digitalis-type drugs
* Patients with insulin-dependent diabetes mellitus whose diabetes has not been stable and controlled for at least the past three months as defined by HbA1C ≥ 10%
* Known drug or alcohol dependency within the past one year period
* Concomitant administration of medications known to affect blood pressure, except medications allowed by the protocol
* Night shift workers who routinely sleep during the daytime and whose work hours include midnight to 4:00 AM
* Patients receiving any investigational therapy within one month of signing the informed consent form. Note that patients who have participated in previous MICARDIS® (telmisartan) studies may participate in this study provided there has been at least one month between discontinuing the previous study and signing the consent for the present study
* Known hypersensitivity to any component of the formulations
* Any clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of trial medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 1998-04; Primary Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in diastolic and systolic blood pressure during the last 6 hours of a 24-hour dosing interval measured by ambulatory blood pressure monitoring (ABPM) | Day 1 and 56 of the open-label period

SECONDARY OUTCOMES:
Changes from baseline in diastolic and systolic blood pressures during other times during 24-hr ABPM profile | Day 1 and 56 of the open-label period
Changes from baseline in seated trough diastolic and systolic blood pressures as measured by manual cuff sphygmomanometer | Baseline (day 27 of the single-blind period), days 1, 14, 28, 56 and 57 of the open-label period
Blood pressure responder rates based on ABPM | day 56 of the open-label period
  24-hour-mean diastolic blood pressure <= 80 mmHg and/or reduction from baseline of at least 10 mmHg or reduction from baseline in 24-hour-mean systolic blood pressure of at least 10 mmHg
Blood pressure responder rates based manual cuff measurements | days 14, 28, 56 and 57 of the open-label period
  24-hour-mean diastolic blood pressure <= 80 mmHg and/or reduction from baseline of at least 10 mmHg or reduction from baseline in 24-hour-mean systolic blood pressure of at least 10 mmHg
Number of patients with adverse events | up to 57 days